CLINICAL TRIAL: NCT06832865
Title: A Phase 2 Study of Elranatamab in Combination With Isatuximab (ELISA) in Relapsed and Refractory Multiple Myeloma
Brief Title: ELISA in Relapsed/Refractory MM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Noopur Raje, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-727
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Relapsed Refractory Multiple Myeloma (RRMM); Relapsed Refractory Multiple Myeloma
Keywords: Prior lines of therapy; relapsed and refractory multiple myeloma; RRMM
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Elranatamab + Isatuximab-irfc (Experimental): Elranatamab will be administered via subcutaneous (SC) injection usually into the abdomen or lower stomach at the following visits during each 28-day cycle:
  * Cycle 1: Days 1, 4, 8, 15, 22
  * Cycles 2-6: Days 1 and 15
  * Cycles 7+: Day 1.
  Isatuximab for SC administration will be administered via subcutaneous (SC) injection usually into the abdomen or lower stomach, using an investigational injector device called the on-body delivery system at the following visits during each 28-day cycle:
  * Cycles 2-6: Days 1 and 15
  * Cycles 7+: Day 1
  This will continue as long as the participant is receiving treatment.
  Interventions: Drug: elranatamab; Drug: Isatuximab SC; Device: Isatuximab SC-OBDS

INTERVENTIONS:
Drug: elranatamab — Subcutaneously injected study drug, usually into the abdomen or lower stomach. Each vial of elranatamab contains a sufficient amount of product to ensure an extractable volume of 1.9 mL at a concentration of 40 mg/mL. The dosing is as follows:
  * Cycle 1 Day 1: 12 mg/0.3 mL
  * Cycle 1 Day 4: 32 mg/0.8 mL
  * Cycle 1 Day 8, 15, 22: 76 mg/1.9 mL
  * Cycles 2-6, Day 1 and 15: 76 mg/1.9 mL
  * Cycles 7+, Day 1: 76 mg/1.9 mL
  Other Names: PF-06863135
Drug: Isatuximab SC — Isatuximab (SAR650984) is an IgG1 derived monoclonal antibody binding selectively the human CD38 membrane protein. Subcutaneously (SC) injected study drug with each vial containing 140 mg/mL (1400 mg/10mL) isatuximab. Isatuximab SC will be injected using the investigational OBDS and in the following doses:
  * Cycles 2-6, Day 1 and 15: 1400 mg/10 mL
  * Cycles 7+ Day 1: 1400 mg/10 mL
  Other Names: SAR650984; Isatuximab irfc
Device: Isatuximab SC-OBDS — The On Body Delivery System (OBDS) also called Isatuximab SC Wearable Injection System, is a sterile, single-use, disposable, elastomeric, user-filled investigational medical device. The OBDD has a reservoir for the drug product (isatuximab). A self-contained, integrated needle (with manual insertion and automatic retraction mechanism) is provided within the OBDS. The OBDS will be used to inject isatuximab each time the participant receives isatuximab in this study. Study drug administration will be done by trained medical professionals in the clinic. The OBDS device will be prepared by the medical professional, placed on the abdomen using the adhesive (sticky) pads that are on the device, the study drug (isatuximab) will be injected, and then the device will be removed.
  Other Names: On Body Delivery System (Device); OBDS; Isatuximab Subcutaneous Injection Device (On Body Delivery System, OBDS); Isatuximab SC Wearable Injection System

SUMMARY:
This is an open-label phase 2 study of elranatamab in combination with isatuximab administered subcutaneously in patients with relapsed and refractory multiple myeloma (RRMM) who have received at least two prior lines of therapy and who have had previous treatment with both immunomodulatory drugs (IMiDs) and a proteasome inhibitor (PI). The subcutaneous injection method of isatuximab administration, including the device used to administer isatuximab, is investigational.

DETAILED DESCRIPTION:
This phase 2, single center, open-label study will enroll 30 patients with relapsed and refractory multiple myeloma (RRMM) who have received at least two prior lines of therapy and who have had previous treatment with both immunomodulatory drugs (IMiDs) and a proteasome inhibitor (PI). Participants with prior therapy with anti-CD38 and anti-B cell maturation antigen (BCMA) target except an anti-BCMA T cell engager (TCE) may be eligible.

This research is being done to see if the study drugs, elranatamab and isatuximab-irfc, reduce the risk of worsening disease and to evaluate the possible risks of the study drugs. Elranatamab is an FDA approved treatment for RRMM. Isatuximab is FDA approved as a treatment option for RRMM when administered intravenously (IV), however isatuximab will be administered as a subcutaneous (SC) infusion (injected under the skin) in this study which is not FDA approved and is investigational. Isatuximab will be administered subcutaneously using an investigational device called the on-body delivery system. The first six patients who complete Cycles 1 and 2 will be assessed for safety and adverse events prior to enrolling all other patients. The research involves screening for eligibility, study treatment and study visits, and follow-up visits. In the beginning (Day 1) of Cycle 1, there may be a 2-8 day inpatient visit so participants can be monitored during their first dose of isatuximab + elranatamab. Participants will receive study treatment until disease progression, unacceptable toxicity, or withdrawal, and will be followed every 3 months for 5 years after their final dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. This study will enroll patients with relapsed and refractory multiple myeloma who have had at least 2 prior lines of therapy including patients who have had previous treatment with both immunomodulatory drugs (IMiDs) and a proteasome inhibitor (PI). Prior therapy with anti-CD38 and anti-B cell maturation antigen (BCMA) target will be permitted except an anti-BCMA T cell engager. Patients cannot be refractory to an anti-CD38 antibody.
* 2. Measurable disease of multiple myeloma as defined by at least one of the following:

  * a. Serum monoclonal protein ≥ 0.5 g/dL. Patients with IgD disease and lower amounts of monoclonal protein may be permitted to enroll with PI approval
  * b. ≥ 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * c. Serum free light chain ≥ 100 mg/L (10 mg/dL) and abnormal serum free kappa to serum free lambda light chain (FLC) ratio (<0.26 or >1.65)
* 3. Age ≥18 years.

  --a. The effects of elranatamab and isatuximab on the developing human fetus are unknown. For this reason and because anti-BCMA bispecific antibodies are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 4 months after the last dose of elranatamab and 5 months after the last dose of isatuximab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* 4. ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* 5. Participants must have adequate organ and marrow function as defined below:

  * a. ANC ≥ 1000/μL. G-CSF is not permitted within 7 days of screening.
  * b. Platelet count ≥ 50,000/µL. Platelet transfusion is not permitted within 7 days of screening.
  * c. Hemoglobin ≥ 8 g/dL. Red blood cell transfusions are permitted to meet eligibility criteria.
  * d. Calculated creatinine clearance of ≥ 30 mL/min by Cockcroft-Gault equation.
  * e. Patient has adequate hepatic function, as evidenced by each of the following:

    * Serum bilirubin values < 2 mg/dL; and
    * Serum aspartate transaminase (ALT) and/or aspartate transaminase (AST) values< 2.5 × the upper limit of normal (ULN) of the institutional laboratory reference range. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval (i.e., total bilirubin <3 mg/dL and normal direct bilirubin).
* 6. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* 7. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* 8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* 1. Patients with active plasma cell leukemia, POEMS syndrome, or amyloidosis are excluded from this trial.
* 2. Stem cell transplant within 12 weeks prior to enrollment, or active GVHD.
* 3. Ongoing Grade ≥2 peripheral sensory or motor neuropathy.
* 4. History of any grade peripheral sensory or motor neuropathy with prior BCMA directed therapy. History of GBS or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.
* 5. Previous treatment with an anti-BCMA bispecific T cell engager.

  --a. Prior treatment with anti-BCMA CAR-T and/or ADC therapy is permitted; however, the participant cannot be refractory to this therapy if it was administered as the last line prior to study enrollment.
* 6. Participants who are receiving any investigational agents currently.
* 7. Participants who have had myeloma therapy or investigational drug within 2 weeks prior to start of treatment or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* 8. Known or suspected hypersensitivity to the study drug or any components of the device (e.g. adhesive which contains acrylic).
* 9. Impaired cardiovascular function or clinically significant cardiovascular diseases, defined as any of the following within 6 months prior to enrollment:

  * a. Acute myocardial infarction, acute coronary syndromes (e.g., unstable angina, coronary artery bypass graft, coronary angioplasty or stenting, pericardial effusion);
  * b. Clinically significant cardiac arrhythmias (e.g., uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * c. Thromboembolic or cerebrovascular events (e.g., transient ischemic attack, cerebrovascular accident, deep vein thrombosis [unless associated with a central venous access complication] or pulmonary embolism);
* 10. Participants with known active HBV, HCV, HIV, or any active, uncontrolled bacterial, fungal, or viral infection. Active infections must be resolved at least 14 days prior to enrollment. Per institutional protocol, HBV DNA testing by PCR is mandatory for subjects at risk for HBV reactivation.
* 11. Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ and or other cancers treated with curative intent.
* 12. Other surgical (including major surgery within past 14 days prior to enrollment) medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* 13. Live attenuated vaccine within 30 days of the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Day 1 to 2 years post-treatment.
  Objective Response will be classified using the International Myeloma Working Group (IMWG) Uniform Response criteria. The rate (ORR) will be calculated using a Simon's two-stage design to test the null hypothesis that the ORR ≤ 0.40 versus the alternative that ORR ≥ 0.60. All patients who receive at least one complete cycle of treatment will be included in a response evaluation. Participants who do not complete cycle 1 (i.e., due to disease progression or who die prior to the end of cycle 1) will not be considered evaluable for response; these participants may be replaced. In the first stage, 22 patients will be accrued. If there are 10 or fewer responses in these 22 patients, the study will be stopped. Otherwise, study will continue to enroll to a total of 30. The null hypothesis will be rejected if 16 or more responses are observed in 30 patients.

SECONDARY OUTCOMES:
Incidence of Drug Related Toxicities | Day 1 to 30 days post-treatment (30 days post last dose). Participants can receive treatment until disease progression, unacceptable toxicity, or withdrawal.
  All participants who receive at least one dose of study treatment will be evaluable for toxicity. CTCAE v5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) CRS and ICANS grading criteria will be used. Adverse events will be summarized on all patients treated. The number of drug related toxicities, and details (categorization and grading) will be described.
Median Progression Free Survival (PFS) | Day 1 through end of follow-up, up to 5 years.
  PFS is defined as the time from start of treatment to disease progression or death from any cause. Patients who have not progressed or died are censored at the date last known progression-free. PFS will be determined according to Kaplan-Meier methodology.
Median Overall Survival (OS) | Day 1 through end of follow-up, up to 5 years.
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive. Median OS will be determined according to Kaplan-Meier methodology.
Rate of Minimal Residual Disease (MRD) status in participants who have achieved very good partial response (VGPR) or complete response (CR) | Screening through 24 months on treatment.
  MRD assessment will be assessed by next generation sequencing via bone marrow aspirate whenever a bone marrow sample is obtained. Those with VGPR or CR (per IMWG) will be included in this assessment. The rate is number of MRD-negative compared to MRD-positive and will be reported at various time points (time of VGPR/CR/sCR (variable, 3-6 months on treatment) and after 12 and 24 months on treatment).
Sustained minimal residual disease (MRD) negative status | Day 1 through 24 months on treatment.
  Rate and number of participants with MRD negative status who have achieved VGPR or CR by IMWG response criteria and have sustained MRD negative status for ≥6 and ≥12 months. MRD assessment will be assessed by next generation sequencing via bone marrow aspirate whenever a bone marrow sample is obtained. Those with VGPR or CR (per IMWG) will be included in this assessment. For patients where CR has been sustained for ≥6 and ≥12 months, MRD evaluation will be repeated to confirm sustained MRD. For patients who are MRD-negative at time of VGPR with persistent VGPR or achieve a CR, MRD evaluation will be repeated to confirm sustained MRD ≥6 and ≥12 months apart. The rate is number of these participants with sustained MRD negative status compared to number without sustained MRD negative status.

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Noopur Raje, MD nraje@mgh.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation